CLINICAL TRIAL: NCT01375075
Title: A Phase 2 Dose Response Study of LY2484595 in Japanese Subjects
Brief Title: A Study of LY2484595 in Japanese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13049; I1V-JE-EIAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Results first posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-03

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — evacetrapib; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 30 milligrams (mg) LY2484595 (Experimental): Administered orally once daily for 12 weeks
  Interventions: Drug: LY2484595; Drug: Placebo
- 100 mg LY2484595 (Experimental): Administered orally once daily for 12 weeks
  Interventions: Drug: LY2484595; Drug: Placebo
- 500 mg LY2484595 (Experimental): Administered orally once daily for 12 weeks
  Interventions: Drug: LY2484595; Drug: Placebo
- Placebo (Placebo Comparator): Administered orally once daily for 12 weeks
  Interventions: Drug: Placebo
- 10 mg Atorvastatin (Active Comparator): Administered orally once daily for 12 weeks
  Interventions: Drug: Placebo; Drug: Atorvastatin
- 100 mg LY2484595 + 10 mg Atorvastatin (Experimental): Administered orally once daily for 12 weeks
  Interventions: Drug: LY2484595; Drug: Placebo; Drug: Atorvastatin

INTERVENTIONS:
Drug: LY2484595 — Administered orally
  Arms: 100 mg LY2484595; 100 mg LY2484595 + 10 mg Atorvastatin; 30 milligrams (mg) LY2484595; 500 mg LY2484595
Drug: Placebo — Administered orally
Drug: Atorvastatin — Administered orally
  Arms: 10 mg Atorvastatin; 100 mg LY2484595 + 10 mg Atorvastatin

SUMMARY:
The purpose of this study is to determine if 12 weeks of treatment with LY2484595 administered as a monotherapy will significantly increase high-density lipoprotein cholesterol (HDL-C) and decrease low-density lipoprotein cholesterol (LDL-C) in Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

Have Low HDL-C or High LDL-C criteria as follows:

Low HDL lipid criteria:

* HDL-C <45 milligrams per deciliter (mg/dL) (men) and <50 mg/dL (women), and
* LDL-C according to Japan Atherosclerosis Society (JAS) guidelines as follows:

  * LDL-C <190 mg/dL (0-1 risk factors)
  * LDL-C <160 mg/dL (2 risk factors)
  * LDL-C <130 mg/dL (3+ risk factors),and
* Fasting Triglycerides (TG) <400 mg/dL

or

High LDL-C lipid criteria:

* HDL-C <100 mg/dL, and
* LDL-C according to JAS guidelines as follows:

  * LDL-C 100-190 mg/dL (0-1 risk factors)
  * LDL-C 100-160 mg/dL (2 risk factors)
  * LDL-C 100-130 mg/dL (3+ risk factors), and
* Fasting TG <400 mg/dL

Note: Subjects with diabetes regarded as 3+ risk factors

* Male subjects: Agree to use a reliable method of birth control during the study (and for 2 weeks following the last dose of study drug)
* Female subjects: 1) Women not of childbearing potential due to surgical sterilization (at least 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy or tubal ligation) confirmed by medical history, or menopause. Menopausal women include women with either a) spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications during the amenorrhea that induced the amenorrhea [for example, oral contraceptives, hormones, gonadotropin releasing hormone, anti-estrogens, selective estrogen receptor modulators (SERMs), or chemotherapy] or b) spontaneous amenorrhea for 6 to 12 months and a follicle-stimulating hormone (FSH) level greater than 40 milli-international units per milliliter (mIU/mL). or, 2) Women of child bearing potential who test negative for pregnancy at the time of enrollment based on a urine or serum pregnancy test and agree to use a reliable method of birth control during the study and for 2 weeks following the last dose of study drug
* Have given informed consent to participate in the study

Exclusion Criteria:

* At screening, are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or unapproved use of a drug or device (other than the investigational product used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated within 90 days prior to screening in any clinical trials of cholesteryl ester transfer protein (CETP) inhibitors (e.g., anacetrapib or dalcetrapib)
* Have completed or withdrawn from this study or have completed or withdrawn from any other study investigating LY2484595
* Are unable, unreliable, and/or unwilling to provide informed consent, make themselves available for the duration of the study, or will not abide by the procedures and study restrictions
* Have recent history of any clinically significant rash, history of any clinically severe drug-related rash, history of a chronic skin disorder (such as psoriasis, eczema or urticaria), history of significant skin hypersensitivities to household or cosmetic products, or allergens per the investigator, or presence of widespread tattoos or other skin condition that limits the assessment for rashes. Subjects who develop any rash during the Diet Lead-in/Washout Phase cannot be randomized
* Have or have had any clinical manifestation of coronary heart disease (CHD), such as stable or unstable angina, acute coronary syndrome, myocardial infarction, or a coronary revascularization procedure including stent placement, symptomatic carotid artery disease or symptomatic peripheral arterial disease. Subjects with a diagnosis of abdominal aortic aneurysm are excluded from this study
* Have systolic blood pressure (SBP) >140 millimeters of mercury (mm Hg) or diastolic blood pressure (DBP) >90 mm Hg as determined by the mean of 3 standardized measurements in the sitting position at randomization
* Have or have had documented hyperaldosteronism
* Have symptoms consistent with moderate or severe heart failure or are receiving treatment for symptomatic congestive heart failure (CHF) or known left ventricular ejection fraction (LVEF) <35%. The absence of LVEF measurement does not prohibit entry into this study
* Have one of the following abnormalities: QTc prolongation [Bazett's corrected QT interval (QTcB)] of >450 msec in male subjects or >470 msec in female subjects, or abnormally wide QRS complexes (resulting from bundle branch blocks, intraventricular conduction delays, or pacemakers) or atrial fibrillation on screening electrocardiogram (ECG), previous history of QTc prolongation with another medication that required discontinuation, congenital long QT syndrome, previous history of ventricular tachycardia or unexplained syncope
* Have family history of long QT syndrome or sudden death likely secondary to ventricular arrhythmia
* Have active hepatobiliary disease, serologic evidence of past or active hepatitis B or C, or past or active gallbladder disease. Subjects who have been diagnosed with Gilbert syndrome or had a cholecystectomy greater than 90 days prior to screening can be included
* Have aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT), alkaline phosphatase (ALP), or total bilirubin >1.5 times the upper limit of normal (ULN)
* Have a history or presence of a chronic muscular or neuromuscular disease including prior rhabdomyolysis or drug-induced myopathy or an unexplained/documented elevation in creatine kinase (CK) ≥3 times the ULN
* Have a history of discontinuation from statin, change of statin, or a dose reduction of statin due to history of hypersensitivity, intolerance or adverse effect. Have a history of increased hepatic enzymes associated with use of an hydroxymethylglutaryl-coenzyme A (HMG-CoA) reductase inhibitor (statin)
* Have a history of hypersensitivity or intolerance to drug preparations containing cholesteryl ester transfer protein (CETP) inhibitors, including but not limited to torcetrapib, anacetrapib, or dalcetrapib
* Have a hemoglobin A1c ≥8.0%; or use, plan to use, or are likely to require insulin during the course of the study. Diabetic subjects on an antidiabetic agent with lipid modifying effects must be on a stable dose for at least 30 days prior to screening
* Have a serum creatinine ≥2 mg/dL, or nephrotic syndrome, end stage renal disease and use renal replacement therapy such as hemodialysis or peritoneal dialysis
* Have hemoglobin <10 grams per deciliter (g/dL) in women and <11 g/dL in men
* Have current uncontrolled active inflammatory condition or infection which in the opinion of the investigator would influence a subject's ability to complete the study
* Have thyroid-stimulating hormone (TSH) levels outside normal reference range. Subjects who are clinically euthyroid, on stable thyroid replacement therapy for 60 days prior to screening, and are anticipated to remain on this dose throughout the trial period are acceptable exceptions to this criterion
* Are women who are lactating
* Have planned or are likely to require major surgery requiring anesthesia or hospitalization during the course of the study
* Have chronic alcohol or drug abuse or dependency
* Are currently under suspicion of having cancer or have had a history of cancer in the past 2 years, with the exception of excised superficial lesions such as basal cell carcinoma and squamous cell carcinoma of the skin
* Have history of human immunodeficiency virus (HIV) infection
* Have any other condition or abnormal laboratory value, which in the opinion of the investigator precludes the subject from providing informed consent
* Plan to use, are likely to require, or unwilling or unable to stop with adequate washout any prescription or over-the-counter (OTC) medication or health foods with the intent to treat serum lipids (LDL-C, HDL-C, triglycerides) including but not limited to these classes of drugs: statin, ezetimibe, bile acid sequestrant, eicosapentaenoic acid (EPA). Subjects taking probucol, fibrate or nicotinic agents within 8 weeks before screening are excluded from the study
* Are currently using, plan to use, or are likely to require during the course of the study systemic corticosteroids; or anabolic agents other than stable doses of estrogen, estrogen/progestin, or testosterone replacement therapy
* Are currently using, plan to use, or are likely to require during the course of the study, more than the occasional use (i.e., once every other week) of stimulant laxatives (e.g., bisacodyl), osmotic laxatives (e.g., milk of magnesia), or castor oil
* Use of any immunosuppressive therapy within 60 days prior to screening or are likely to require immunosuppressive therapy during the course of the study
* Have received treatment within 30 days prior to the time of study entry with any drug or drugs that have not received regulatory approval for any indication
* Have plans to adopt diets with aggressive carbohydrate restrictions for weight loss. Currently use, have used within 60 days prior to screening, or plan to use during the trial period prescriptions or OTC formulations intended for weight loss
* Are currently using, have used within 60 days prior to screening, plan to use, or are likely to require during the course of the study, drugs or foods that are inducers (including rifampin and carbamazepine) or moderate or strong inhibitors of cytochrome P450 3A (including, ketoconazole, erythromycin and grapefruit juice); or strong inhibitors of the organic anion transporter polypeptide 1B1 (OATP1B1) transporter (including cyclosporine and rifampin). The drugs used in topical preparations are acceptable

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- Japan (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, participants stopped lipid-related concomitant medications and started a diet therapy in accordance with the Japan Atherosclerosis Society guidelines for diagnosis and prevention of atherosclerotic cardiovascular disease.
Groups:
- 30 mg LY2484595: The following were administered orally once daily for 12 weeks:
  Placebo (LY2484595): 4 tablets
  Placebo (Atorvastatin): 1 capsule
  LY2484595: A single 30-milligram (mg) tablet
- 100 mg LY2484595: The following were administered orally once daily for 12 weeks:
  Placebo (LY2484595): 4 tablets
  Placebo (Atorvastatin): 1 capsule
  LY2484595: A single 100-mg tablet
- 500 mg LY2484595: The following were administered orally once daily for 12 weeks:
  Placebo (Atorvastatin): 1 capsule
  LY2484595: five 100-mg tablets
- Placebo: The following were administered orally once daily for 12 weeks:
  Placebo (LY2484595): 5 tablets
  Placebo (Atorvastatin): 1 capsule
- 10 mg Atorvastatin: The following were administered orally once daily for 12 weeks:
  Atorvastatin: A single 10-mg capsule
  Placebo (LY2484595): 5 tablets
- 100 mg LY2484595 + 10 mg Atorvastatin: The following were administered orally once daily for 12 weeks:
  Atorvastatin: A single 10-mg capsule
  LY2484595: A single 100-mg tablet
  Placebo (LY2484595): 4 tablets
Period: Overall Study
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Started | 27 | 28 | 27 | 28 | 27 | 28
Received at Least One Dose of Study Drug | 27 | 28 | 27 | 28 | 27 | 28
Completed | 26 | 27 | 24 | 27 | 27 | 25
Not Completed | 1 | 1 | 3 | 1 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 3 | 1 | 0 | 1
Not completed — Entry Criterion Not Met | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 30 mg LY2484595: The following were administered orally once daily for 12 weeks:
  Placebo (LY2484595): 4 tablets
  Placebo (Atorvastatin): 1 capsule LY2484595: A single 30-mg tablet
- Total: Total of all reporting groups
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin | Total
Number analyzed (Participants) | 27 | 28 | 27 | 28 | 27 | 28 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (10.95) | 47.6 (11.94) | 49.4 (8.10) | 50.3 (9.63) | 49.4 (8.76) | 50.0 (10.01) | 49.2 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 9 | 10 | 8 | 10 | 55
  Male | 19 | 18 | 18 | 18 | 19 | 18 | 110
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 27 | 28 | 27 | 28 | 27 | 28 | 165
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 27 | 28 | 27 | 28 | 27 | 28 | 165
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 68.5 (14.04) | 65.9 (11.58) | 68.5 (15.71) | 69.3 (13.51) | 67.4 (12.77) | 70.3 (18.33) | 68.3 (14.34)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 165.1 (9.48) | 165.4 (9.95) | 166.5 (9.27) | 165.6 (8.56) | 166.7 (6.76) | 165.2 (8.34) | 165.7 (8.68)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m²)] | 24.9 (3.38) | 24.0 (3.15) | 24.5 (4.10) | 25.1 (3.70) | 24.1 (3.35) | 25.5 (5.49) | 24.7 (3.93)
Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 143.9 (24.02) | 143.6 (23.05) | 142.6 (30.16) | 140.1 (27.37) | 134.3 (31.78) | 139.6 (19.84) | 140.7 (26.12)
High-Density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 50.2 (12.88) | 52.1 (16.15) | 49.2 (11.41) | 50.7 (14.39) | 48.9 (13.70) | 51.7 (14.47) | 50.5 (13.77)
Fasting Triglycerides (TG) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 156.1 (74.31) | 133.1 (64.75) | 145.4 (79.14) | 138.9 (64.56) | 143.1 (60.02) | 144.3 (75.32) | 143.4 (69.27)
Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] | 118.8 (11.75) | 117.7 (12.41) | 118.4 (12.61) | 119.5 (11.67) | 119.6 (9.82) | 116.9 (13.31) | 118.5 (11.84)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] | 73.7 (7.32) | 74.0 (9.57) | 74.3 (9.77) | 75.1 (7.32) | 75.4 (7.58) | 71.8 (8.52) | 74.0 (8.37)
Pulse Rate [Mean (Standard Deviation); unit: beats per minute (bpm)] | 68.4 (8.90) | 67.7 (7.45) | 68.2 (10.41) | 67.3 (11.15) | 68.4 (8.14) | 72.4 (8.90) | 68.8 (9.26)

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) and Low Density Lipoprotein Cholesterol (LDL-C) With LY2484595 in Combination With Atorvastatin
Description: Percent change from baseline = 100*(post-baseline assessment - baseline assessment)/baseline assessment. An increase in the percent change from baseline represented an improvement for HDL-C and a decrease in the percent change from baseline represents an improvement for LDL-C. LS mean was adjusted for baseline value of the variable analyzed.
Time Frame: Baseline, Weeks 2, 4, and 8
Population: All randomized participants who took at least 1 dose of double-blind study medication, had a baseline and at least 1 post-baseline HDL-C measurement (mITT population), and had at least 1 post-baseline value of the response variable for the specified time frame.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 27 | 27 | 27 | 28 | 27 | 28
percent change
  HDL-C, Week 2 | 75.30 (6.44) | 108.21 (6.45) | 122.60 (6.44) | -0.73 (6.32) | 8.85 (6.45) | 101.45 (6.33)
  HDL-C, Week 4: number analyzed (Participants) | 27 | 27 | 25 | 27 | 27 | 28
  HDL-C, Week 4 | 77.94 (7.62) | 122.68 (7.63) | 147.22 (7.72) | 2.09 (7.53) | 10.87 (7.62) | 117.04 (7.49)
  HDL-C, Week 8: number analyzed (Participants) | 26 | 27 | 24 | 27 | 27 | 25
  HDL-C, Week 8 | 78.65 (7.95) | 130.69 (7.91) | 169.05 (8.08) | 5.19 (7.82) | 12.98 (7.91) | 116.64 (7.90)
  LDL-C, Week 2 | -17.46 (3.13) | -27.50 (3.14) | -33.19 (3.13) | -2.14 (3.07) | -38.29 (3.14) | -55.74 (3.04)
  LDL-C, Week 4: number analyzed (Participants) | 27 | 27 | 25 | 27 | 27 | 28
  LDL-C, Week 4 | -13.32 (3.14) | -24.43 (3.14) | -29.25 (3.18) | 2.84 (3.10) | -42.23 (3.15) | -52.62 (3.08)
  LDL-C, Week 8: number analyzed (Participants) | 26 | 27 | 24 | 27 | 27 | 25
  LDL-C, Week 8 | -12.50 (3.39) | -23.56 (3.37) | -25.48 (3.45) | 0.24 (3.33) | -38.97 (3.38) | -51.23 (3.38)
Statistical Analysis 1: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in HDL-C at Week 2; Treatment, visit, and treatment by visit interaction were included in the model as fixed effects, baseline measurement as covariate; LS Mean Difference = 92.61, 90% CI 2-sided [77.65 to 107.57], Standard Error of Mean 9.04
Statistical Analysis 2: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in HDL-C at Week 4; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 106.17, 90% CI 2-sided [88.47 to 123.87], Standard Error of Mean 10.69
Statistical Analysis 3: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in HDL-C at Week 8; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 103.66, 90% CI 2-sided [85.14 to 122.17], Standard Error of Mean 11.18
Statistical Analysis 4: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in LDL-C at Week 2; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -17.46, 90% CI 2-sided [-24.73 to -10.19], Standard Error of Mean 4.39
Statistical Analysis 5: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis — The P-value is for percent change from baseline in LDL-C at Week 4; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -10.39, 90% CI 2-sided [-17.67 to -3.11], Standard Error of Mean 4.40
Statistical Analysis 6: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — The P-value is for percent change from baseline in LDL-C at Week 8; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -12.26, 90% CI 2-sided [-20.17 to -4.36], Standard Error of Mean 4.77

2. Secondary Outcome: Pharmacokinetics - Area Under the Curve (AUC) of LY2484595 and Atorvastatin
Time Frame: Weeks 2, 4, 8, 12 (predose and postdose), and Week 16
Population: Participants who were administered LY2484595 or LY2484595 + Atorvastatin and had evaluable pharmacokinetic (PK) samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- 30 mg LY2484595: The following were administered orally once daily for 12 weeks:
  Placebo: 4 tablets and 1 capsule
  LY2484595: A single 30-milligram (mg) tablet
- 100 mg LY2484595: The following were administered orally once daily for 12 weeks:
  Placebo: 4 tablets and 1 capsule
  LY2484595: A single 100-mg tablet
- 100 mg LY2484595 + 10 mg Atorvastatin: The following were administered orally once daily for 12 weeks:
  Atorvastatin: A single 10-mg capsule
  Placebo: 4 tablets
  LY2484595: A single 100-mg tablet
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 27 | 27 | 26 | 27
nanograms*hours per milliliter (ng*h/mL) | 3110 (32) | 8690 (44) | 29400 (42) | 8080 (47)

3. Secondary Outcome: The Number and Severity of Episodes of Rashes at Any Time From Baseline Through Week 12
Description: All rash cases were adjudicated by a central dermatologist blinded to treatment assignment according to a study-specific Clinical Events Committee (CEC) charter. Rash events were assessed according to clinical relevance (severity). Categories included high risk, low risk, not a relevant dermatosis, or insufficient documentation for determination. High risk rashes included anaphylaxis, toxic epidermal necrolysis, Stevens Johnson Syndrome, Drug Reaction with Eosinophilia and System Symptoms (DRESS), urticaria/angioedema, vasculitis, erythroderma, and lupus-like reaction. All other rashes were considered low risk or not a relevant dermatosis per the Investigator's clinical opinion. A participant could be reported in multiple categories.
Time Frame: Baseline through Week 12
Population: All randomized participants who took at least 1 dose of double-blind study medication intent-to-treat (ITT) population.
Measure: Number; unit: events
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 27 | 28 | 27 | 28 | 27 | 28
events
  Low risk | 0 | 0 | 1 | 0 | 0 | 1
  High risk | 0 | 0 | 1 | 0 | 0 | 0
  Not a relevant dermatosis | 0 | 0 | 0 | 1 | 0 | 1
  Insufficient documentation for determination | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline to 12 Weeks in Blood Pressure
Description: Blood pressure reported as systolic blood pressure (SBP) and diastolic blood pressure (DBP).
  LS mean was adjusted for baseline value of the variable analyzed.
Time Frame: Baseline and Week 12
Population: All randomized participants who took at least 1 dose of double-blind study medication (ITT population) and had a baseline and at least 1 post-baseline value of the response variable.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mm Hg)
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 26 | 27 | 24 | 27 | 27 | 25
millimeters of mercury (mm Hg)
  SBP | 2.35 (1.78) | 1.44 (1.76) | 4.51 (1.84) | -1.39 (1.75) | 2.59 (1.76) | 2.04 (1.80)
  DBP | 1.46 (1.07) | 0.02 (1.05) | 2.51 (1.10) | 0.68 (1.05) | 1.49 (1.05) | 0.51 (1.08)
Statistical Analysis 1: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.136, Mixed Models Analysis — The P-value is for change from baseline in SBP at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 3.74, 90% CI 2-sided [-0.39 to 7.88], Standard Error of Mean 2.50
Statistical Analysis 2: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.257, Mixed Models Analysis — The P-value is for change from baseline in SBP at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.83, 90% CI 2-sided [-1.28 to 6.94], Standard Error of Mean 2.48
Statistical Analysis 3: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.021, Mixed Models Analysis — The P-value is for change from baseline in SBP at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 5.90, 90% CI 2-sided [1.70 to 10.10], Standard Error of Mean 2.54
Statistical Analysis 4: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.829, Mixed Models Analysis — The P-value is for change from baseline in SBP at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.54, 90% CI 2-sided [-4.71 to 3.62], Standard Error of Mean 2.52
Statistical Analysis 5: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.603, Mixed Models Analysis — The P-value is for change from baseline in DBP at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.78, 90% CI 2-sided [-1.69 to 3.24], Standard Error of Mean 1.50
Statistical Analysis 6: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.656, Mixed Models Analysis — The P-value is for change from baseline in DBP at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.66, 90% CI 2-sided [-3.11 to 1.78], Standard Error of Mean 1.48
Statistical Analysis 7: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.228, Mixed Models Analysis — The P-value is for change from baseline in DBP at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.83, 90% CI 2-sided [-0.67 to 4.34], Standard Error of Mean 1.52
Statistical Analysis 8: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.516, Mixed Models Analysis — The P-value is for change from baseline in DBP at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.98, 90% CI 2-sided [-3.47 to 1.51], Standard Error of Mean 1.51

5. Secondary Outcome: Change From Baseline to 12 Weeks in Aldosterone
Description: LS mean was adjusted for baseline value of the variable analyzed.
Time Frame: Baseline and Week 12
Population: All randomized participants who took at least 1 dose of double-blind study medication (ITT population) and had a baseline and at least 1 post-baseline aldosterone measurement.
Measure: Least Squares Mean (Standard Error); unit: nanograms per deciliter (ng/dL)
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 25 | 25 | 21 | 25 | 25 | 24
nanograms per deciliter (ng/dL) | -0.40 (0.79) | 0.37 (0.79) | 0.59 (0.84) | 0.33 (0.79) | 0.95 (0.79) | 0.62 (0.79)
Statistical Analysis 1: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.513, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.73, 90% CI 2-sided [-2.57 to 1.11], Standard Error of Mean 1.11
Statistical Analysis 2: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.970, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.04, 90% CI 2-sided [-1.82 to 1.90], Standard Error of Mean 1.12
Statistical Analysis 3: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.824, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.26, 90% CI 2-sided [-1.66 to 2.17], Standard Error of Mean 1.16
Statistical Analysis 4: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.769, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.33, 90% CI 2-sided [-2.18 to 1.52], Standard Error of Mean 1.12

6. Secondary Outcome: Change From Baseline to 12 Weeks in Plasma Renin Activity
Description: LS mean was adjusted for baseline value of the variable analyzed.
Time Frame: Baseline and Week 12
Population: All randomized participants who took at least 1 dose of double-blind study medication (ITT population) and had a baseline and at least 1 post-baseline plasma renin activity measurement.
Measure: Least Squares Mean (Standard Error); unit: nanograms per milliliter per hour
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 24 | 24 | 24 | 26 | 26 | 24
nanograms per milliliter per hour | -0.32 (0.23) | 0.01 (0.24) | -0.21 (0.23) | -0.21 (0.23) | -0.01 (0.23) | -0.43 (0.23)
Statistical Analysis 1: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.735, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.11, 90% CI 2-sided [-0.65 to 0.43], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.503, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.22, 90% CI 2-sided [-0.32 to 0.76], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.988, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.00, 90% CI 2-sided [-0.53 to 0.54], Standard Error of Mean 0.33
Statistical Analysis 4: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.207, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.41, 90% CI 2-sided [-0.95 to 0.13], Standard Error of Mean 0.32

7. Secondary Outcome: Change From Baseline to 12 Weeks in Serum Sodium
Description: LS mean was adjusted for baseline value of the variable analyzed.
Time Frame: Baseline and Week 12
Population: All randomized participants who took at least 1 dose of double-blind study medication (ITT population) and had a baseline and at least 1 post-baseline serum sodium measurement.
Measure: Least Squares Mean (Standard Error); unit: milliequivalents per liter (mEq/L)
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 26 | 27 | 24 | 27 | 27 | 25
milliequivalents per liter (mEq/L) | -0.18 (0.31) | -0.32 (0.30) | -0.07 (0.32) | -0.32 (0.30) | 0.35 (0.30) | 0.53 (0.31)
Statistical Analysis 1: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.756, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.13, 90% CI 2-sided [-0.57 to 0.84], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.990, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.01, 90% CI 2-sided [-0.71 to 0.70], Standard Error of Mean 0.43
Statistical Analysis 3: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.565, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.25, 90% CI 2-sided [-0.47 to 0.97], Standard Error of Mean 0.44
Statistical Analysis 4: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.678, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.18, 90% CI 2-sided [-0.53 to 0.89], Standard Error of Mean 0.43

8. Secondary Outcome: Change From Baseline to 12 Weeks in Serum Bicarbonate
Description: LS mean was adjusted for baseline value of the variable analyzed.
Time Frame: Baseline and Week 12
Population: All randomized participants who took at least 1 dose of double-blind study medication (ITT population) and had a baseline and at least 1 post-baseline serum bicarbonate measurement.
Measure: Least Squares Mean (Standard Error); unit: milliequivalents per liter (mEq/L)
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 26 | 27 | 24 | 27 | 27 | 25
milliequivalents per liter (mEq/L) | 0.63 (0.43) | 0.62 (0.43) | 0.62 (0.45) | 0.52 (0.43) | 0.62 (0.43) | 1.23 (0.44)
Statistical Analysis 1: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.856, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.11, 90% CI 2-sided [-0.90 to 1.12], Standard Error of Mean 0.61
Statistical Analysis 2: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.869, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.10, 90% CI 2-sided [-0.90 to 1.10], Standard Error of Mean 0.61
Statistical Analysis 3: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.869, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.10, 90% CI 2-sided [-0.92 to 1.13], Standard Error of Mean 0.62
Statistical Analysis 4: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.317, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.61, 90% CI 2-sided [-0.40 to 1.63], Standard Error of Mean 0.61

9. Secondary Outcome: Number of Myopathy and Liver Injury Events
Description: Myopathy events were considered muscle-related treatment emergent adverse events (TEAEs) and liver injury events were considered hepatic disorder-related TEAEs reported per Medical Dictionary for Regulatory Activities (MedDRA). An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. TEAEs were newly occurring AEs or AEs worsening after first dose.
Time Frame: Baseline through Week 12
Population: All randomized participants who took at least 1 dose of double-blind study medication (ITT population).
Measure: Number; unit: events
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 27 | 28 | 27 | 28 | 27 | 28
events
  Blood creatine phosphokinase increased | 0 | 1 | 0 | 0 | 1 | 0
  Myalgia | 0 | 1 | 0 | 0 | 1 | 0
  Hepatic function abnormal | 1 | 0 | 1 | 0 | 1 | 2
  Gamma-glutamyltransferase increased | 0 | 1 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 0 | 0 | 0 | 1 | 0 | 0

10. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Highly-Sensitive C-Reactive Protein (hsCRP)
Description: LS mean was adjusted for baseline value of the variable analyzed.
Time Frame: Baseline and Week 12
Population: All randomized participants who took at least 1 dose of double-blind study medication, had a baseline and at least 1 post-baseline HDL-C measurement (mITT population), and had at least 1 post-baseline hsCRP measurement.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 27 | 27 | 27 | 28 | 27 | 28
milligrams per deciliter (mg/dL) | -0.03 (0.10) | 0.00 (0.10) | 0.13 (0.09) | -0.01 (0.09) | -0.03 (0.10) | 0.15 (0.09)
Statistical Analysis 1: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.888, ANCOVA; Treatment was included in the model as fixed effects, baseline hsCRP as covariate; LS Mean Difference = -0.02, 90% CI 2-sided [-0.24 to 0.20], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.939, ANCOVA; Treatment was included in the model as fixed effects, baseline hsCRP as covariate; LS Mean Difference = 0.01, 90% CI 2-sided [-0.21 to 0.23], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p = 0.296, ANCOVA; Treatment was included in the model as fixed effects, baseline hsCRP as covariate; LS Mean Difference = 0.14, 90% CI 2-sided [-0.08 to 0.36], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.181, ANCOVA; Treatment was included in the model as fixed effects, baseline hsCRP as covariate; LS Mean Difference = 0.18, 90% CI 2-sided [-0.04 to 0.40], Standard Error of Mean 0.13

11. Secondary Outcome: Percent Change From Baseline in Plasma Cholesteryl Ester Transfer Protein (CETP) Activity
Description: Plasma CETP activity assay employed a fluorometric method to determine the CETP transfer activity. Percent change from baseline = 100*(post-baseline assessment - baseline assessment)/baseline assessment. An increase in the percent change from baseline represented an improvement. LS mean was adjusted for baseline value of the variable analyzed.
Time Frame: Baseline, Weeks 4, 8, and 12
Population: All randomized participants who took at least 1 dose of double-blind study medication, had a baseline and at least 1 post-baseline HDL-C measurement (mITT population), and had at least 1 post-baseline CETP activity measurement.
Measure: Least Squares Mean (Standard Error); unit: percent change in CETP activity
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 27 | 26 | 25 | 27 | 27 | 27
percent change in CETP activity
  4 Weeks | -41.62 (4.23) | -75.26 (4.30) | -89.14 (4.38) | 1.67 (4.22) | -1.33 (4.22) | -68.58 (4.21)
  8 Weeks: number analyzed (Participants) | 25 | 26 | 24 | 27 | 27 | 23
  8 Weeks | -39.91 (4.47) | -76.23 (4.40) | -90.97 (4.57) | 2.70 (4.32) | -4.89 (4.32) | -79.90 (4.60)
  12 Weeks: number analyzed (Participants) | 26 | 26 | 24 | 27 | 26 | 23
  12 Weeks | -41.07 (3.57) | -73.86 (3.55) | -85.30 (3.69) | 9.22 (3.49) | -5.69 (3.54) | -73.38 (3.74)
Statistical Analysis 1: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 4; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -43.29, 90% CI 2-sided [-53.16 to -33.41], Standard Error of Mean 5.97
Statistical Analysis 2: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 4; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -76.93, 90% CI 2-sided [-86.89 to -66.97], Standard Error of Mean 6.02
Statistical Analysis 3: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 4; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -90.81, 90% CI 2-sided [-100.87 to -80.75], Standard Error of Mean 6.08
Statistical Analysis 4: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 4; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -67.25, 90% CI 2-sided [-77.12 to -57.39], Standard Error of Mean 5.96
Statistical Analysis 5: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 8; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -42.60, 90% CI 2-sided [-52.88 to -32.33], Standard Error of Mean 6.21
Statistical Analysis 6: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 8; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -78.93, 90% CI 2-sided [-89.15 to -68.71], Standard Error of Mean 6.17
Statistical Analysis 7: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 8; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -93.67, 90% CI 2-sided [-104.08 to -83.26], Standard Error of Mean 6.29
Statistical Analysis 8: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 8; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -75.01, 90% CI 2-sided [-85.46 to -64.57], Standard Error of Mean 6.31
Statistical Analysis 9: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -50.28, 90% CI 2-sided [-58.53 to -42.04], Standard Error of Mean 4.98
Statistical Analysis 10: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -83.07, 90% CI 2-sided [-91.32 to -74.83], Standard Error of Mean 4.98
Statistical Analysis 11: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -94.51, 90% CI 2-sided [-102.92 to -86.10], Standard Error of Mean 5.08
Statistical Analysis 12: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in plasma CETP activity at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -67.68, 90% CI 2-sided [-76.20 to -59.16], Standard Error of Mean 5.15

12. Secondary Outcome: Change From Baseline in Plasma CETP Mass
Description: Plasma CETP mass assay was a solid-phase enzyme-linked immunosorbent assay (ELISA) designated to measure human CETP mass which employed the quantitative enzyme immunoassay principle. An increase in plasma CETP mass represented an improvement. LS mean was adjusted for baseline value of the variable analyzed.
Time Frame: Baseline, Weeks 4, 8, and 12
Population: All randomized participants who took at least 1 dose of double-blind study medication, had a baseline and at least 1 post-baseline HDL-C measurement (mITT population), and had at least 1 post-baseline CETP mass measurement.
Measure: Least Squares Mean (Standard Error); unit: micrograms per milliliter (µg/mL)
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 27 | 27 | 25 | 27 | 27 | 28
micrograms per milliliter (µg/mL)
  4 weeks | 1.88 (0.18) | 3.14 (0.18) | 3.54 (0.18) | 0.08 (0.18) | -0.28 (0.18) | 1.94 (0.17)
  8 weeks: number analyzed (Participants) | 26 | 27 | 24 | 27 | 27 | 25
  8 weeks | 1.98 (0.21) | 3.09 (0.21) | 4.02 (0.22) | 0.10 (0.21) | -0.21 (0.21) | 1.83 (0.21)
  12 weeks: number analyzed (Participants) | 26 | 27 | 24 | 27 | 27 | 25
  12 weeks | 1.95 (0.21) | 2.96 (0.21) | 3.36 (0.22) | 0.13 (0.21) | -0.19 (0.21) | 1.95 (0.21)
Statistical Analysis 1: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 4; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.80, 90% CI 2-sided [1.38 to 2.21], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 4; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 3.06, 90% CI 2-sided [2.65 to 3.48], Standard Error of Mean 0.25
Statistical Analysis 3: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 4; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 3.46, 90% CI 2-sided [3.04 to 3.88], Standard Error of Mean 0.25
Statistical Analysis 4: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 4; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.22, 90% CI 2-sided [1.81 to 2.63], Standard Error of Mean 0.25
Statistical Analysis 5: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 8; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.88, 90% CI 2-sided [1.40 to 2.36], Standard Error of Mean 0.29
Statistical Analysis 6: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 8; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.99, 90% CI 2-sided [2.51 to 3.47], Standard Error of Mean 0.29
Statistical Analysis 7: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 8; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 3.92, 90% CI 2-sided [3.42 to 4.41], Standard Error of Mean 0.30
Statistical Analysis 8: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 8; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.04, 90% CI 2-sided [1.56 to 2.52], Standard Error of Mean 0.29
Statistical Analysis 9: Comparison: 30 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.82, 90% CI 2-sided [1.34 to 2.31], Standard Error of Mean 0.29
Statistical Analysis 10: Comparison: 100 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.83, 90% CI 2-sided [2.34 to 3.31], Standard Error of Mean 0.29
Statistical Analysis 11: Comparison: 500 mg LY2484595 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 3.24, 90% CI 2-sided [2.74 to 3.73], Standard Error of Mean 0.30
Statistical Analysis 12: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for change from baseline in plasma CETP mass at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.14, 90% CI 2-sided [1.65 to 2.63], Standard Error of Mean 0.29

13. Primary Outcome: Percent Change From Baseline to 12 Weeks in High Density Lipoprotein Cholesterol (HDL-C) and Low Density Lipoprotein Cholesterol (LDL-C) With LY2484595 and Placebo
Description: Percent change from baseline = 100*(post-baseline assessment - baseline assessment)/baseline assessment. Higher values in the percent change from baseline represented an improvement for HDL-C and lower values in the percent change from baseline represented an improvement for LDL-C. Least Squares (LS) mean was adjusted for baseline value of the variable analyzed.
Time Frame: Baseline and Week 12
Population: All randomized participants who took at least 1 dose of double-blind study medication, had a baseline and at least 1 post-baseline HDL-C measurement [modified intent-to-treat (mITT) population], and also completed the Week 12 visit.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Number analyzed (Participants) | 26 | 27 | 24 | 27 | 27 | 25
percent change
  HDL-C | 82.22 (8.97) | 123.35 (8.92) | 143.56 (9.16) | 8.00 (8.83) | 17.35 (8.91) | 120.60 (8.95)
  LDL-C | -14.23 (3.46) | -22.13 (3.43) | -20.95 (3.55) | 1.24 (3.40) | -37.66 (3.44) | -52.29 (3.47)
Statistical Analysis 1: Comparison: 30 mg LY2484595 vs Placebo; Comparisons between LY2484595 and Placebo were the primary focus for this endpoint; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in HDL-C at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 74.23, 90% CI 2-sided [53.38 to 95.07], Standard Error of Mean 12.59
Statistical Analysis 2: Comparison: 100 mg LY2484595 vs Placebo; Comparisons between LY2484595 and Placebo were the primary focus for this endpoint; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in HDL-C at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 115.36, 90% CI 2-sided [94.58 to 136.14], Standard Error of Mean 12.55
Statistical Analysis 3: Comparison: 500 mg LY2484595 vs Placebo; Comparisons between LY2484595 and Placebo were the primary focus for this endpoint; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in HDL-C at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 135.57, 90% CI 2-sided [114.50 to 156.63], Standard Error of Mean 12.72
Statistical Analysis 4: Comparison: 30 mg LY2484595 vs Placebo; Comparisons between LY2484595 and Placebo were the primary focus for this endpoint; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — The P-value is for percent change from baseline in LDL-C at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -15.47, 90% CI 2-sided [-23.50 to -7.43], Standard Error of Mean 4.85
Statistical Analysis 5: Comparison: 100 mg LY2484595 vs Placebo; Comparisons between LY2484595 and Placebo were the primary focus for this endpoint; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in LDL-C at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -23.37, 90% CI 2-sided [-31.37 to -15.38], Standard Error of Mean 4.83
Statistical Analysis 6: Comparison: 500 mg LY2484595 vs Placebo; Comparisons between LY2484595 and Placebo were the primary focus for this endpoint; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in LDL-C at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -22.19, 90% CI 2-sided [-30.32 to -14.06], Standard Error of Mean 4.91
Statistical Analysis 7: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — The P-value is for percent change from baseline in HDL-C at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 103.25, 90% CI 2-sided [82.32 to 124.18], Standard Error of Mean 12.64
Statistical Analysis 8: Comparison: 10 mg Atorvastatin vs 100 mg LY2484595 + 10 mg Atorvastatin; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — The P-value is for percent change from baseline in LDL-C at Week 12; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -14.63, 90% CI 2-sided [-22.72 to -6.55], Standard Error of Mean 4.88

ADVERSE EVENTS:
Arm/Group | 30 mg LY2484595 | 100 mg LY2484595 | 500 mg LY2484595 | Placebo | 10 mg Atorvastatin | 100 mg LY2484595 + 10 mg Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 1/27 | 1/28 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 12/27 | 12/28 | 10/27 | 8/28 | 10/27 | 10/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 mg LY2484595 (N=27) | 100 mg LY2484595 (N=28) | 500 mg LY2484595 (N=27) | Placebo (N=28) | 10 mg Atorvastatin (N=27) | 100 mg LY2484595 + 10 mg Atorvastatin (N=28)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 mg LY2484595 (N=27) | 100 mg LY2484595 (N=28) | 500 mg LY2484595 (N=27) | Placebo (N=28) | 10 mg Atorvastatin (N=27) | 100 mg LY2484595 + 10 mg Atorvastatin (N=28)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periproctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (4) | 6 (6) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days